CLINICAL TRIAL: NCT00084617
Title: Phase II Study of Oxaliplatin, Irinotecan, and Capecitabine in Advanced Gastric/Gastroesophageal Junction Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03010; CASE 1203; CDR0000365464; U01CA062502 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2013-07

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Irinotecan; Capecitabine

ARMS (1):
- Treatment (oxaliplatin, irinotecan, capecitabine) (Experimental): Patients receive oxaliplatin IV over 2 hours and irinotecan IV over 30 minutes on days 1, 8, 15, and 22 and oral capecitabine twice daily on days 1-5, 8-12, 15-19, and 22-26. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: irinotecan hydrochloride; Drug: capecitabine

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: capecitabine — Given orally
  Other Names: CAPE; Ro 09-1978/000; Xeloda

SUMMARY:
Drugs used in chemotherapy, such as oxaliplatin, irinotecan, and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one chemotherapy drug may kill more tumor cells. This phase II trial is studying how well giving oxaliplatin together with irinotecan and capecitabine works in treating patients with metastatic or inoperable locally advanced gastric cancer or gastroesophageal junction adenocarcinoma (cancer).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the total response rate of the oxaliplatin, irinotecan and capecitabine drug combination in advanced gastric/esophageal junction carcinoma.

II. To assess the duration of total responses of the oxaliplatin, irinotecan and capecitabine drug combination in advanced gastric/esophageal junction carcinoma.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin IV over 2 hours and irinotecan IV over 30 minutes on days 1, 8, 15, and 22 and oral capecitabine twice daily on days 1-5, 8-12, 15-19, and 22-26. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 40-80 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction. Patients must have metastatic or inoperable locally advanced disease; GE Junction tumor location should be documented in the patient's medical record chart using the Siewert classification below:

  * Type I: Adenocarcinoma of the distal esophagus which usually arises from an area with specialized intestinal metaplasia of the esophagus and which may infiltrate the GE junction from above Type II: True carcinoma of the cardia arising from the cardiac epithelium or short segments with intestinal metaplasia at the GE junction Type III: Subcardial gastric carcinoma which infiltrates the GE junction and distal esophagus from below
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* No prior chemotherapy for metastatic or recurrent disease is allowed; one course of neoadjuvant chemotherapy and/or adjuvant chemotherapy with or without radiation therapy as primary treatment is acceptable; at least 4 weeks must have elapsed since prior radiation therapy; patients must have been off previous anti-cancer therapy for at least 4 weeks
* Life expectancy of >= 12 weeks
* ECOG performance status 0-2
* Hemoglobin >= 9.5 g/dL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 mg/dL
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of oxaliplatin, irinotecan, and capecitabine on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because these drugs are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; patients should have no greater than grade 2 neuropathy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, irinotecan and capecitabine
* Patients with NYHA classification III or IV heart disease are ineligible
* Patients must not have a known hypersensitivity to 5-fluorouracil
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the study drugs have the potential to cause teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drugs, breastfeeding should be discontinued if the mother is treated with oxaliplatin, irinotecan or capecitabine
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with the study drugs; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients who are unable to take oral medications are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-03; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Brell, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center single treatment arm study involving four sites. Patients were recruited February 2004 through February 2007.
Period: Overall Study
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Started | 39
Completed | 30
Not Completed | 9
Not completed — Withdrawal by Subject | 7
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 57.8 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Response Rates (RR) in Metastatic Gastric/GE Junction Tumors
Description: Response is defined as the number of patients with a CR (Complete Response) or PR (Partial Response) per Response Evaluation Criteria in Solid Tumor (RECIST criteria). Possible evaluations include: CR: Disappearance of all target lesions. PR: At least a 30% decrease in the size of target lesions. Progressive Disease (PD): At least a 20% increase in the size of the target lesions or appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage or increase of target lesions.
Time Frame: at 12 weeks (after 2 cycles of treatment)
Population: Patients that completed at least 2 cycles of treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Number analyzed (Participants) | 30
participants
  Complete Response (CR) | 2
  Partial Response (PR) | 9
  Progressive Disease (PD) | 3
  Stable Disease (SD) | 16

2. Secondary Outcome: Complete Response (CR) and Partial Response (PR) Duration
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: at 40 months from study activation
Population: Patients that achieved either a CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Number analyzed (Participants) | 11
months | 5.95 [2.07 to 10.55]

3. Secondary Outcome: Overall Survival
Description: Length of time patients survived after treatment
Time Frame: at 40 months from study activation
Population: All patients enrolled in study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Number analyzed (Participants) | 39
months | 8.98 [6.85 to 13.31]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed while patients were on study for up to 4 years
Arm/Group | Treatment (Oxaliplatin, Irinotecan, Capecitabine)
Serious Adverse Events (participants affected / at risk) | 7/39
Other Adverse Events (participants affected / at risk) | 35/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Oxaliplatin, Irinotecan, Capecitabine) (N=39)
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 1
Seizure (Nervous system disorders) | 1
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Perforation, GI - Esophagus (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Oxaliplatin, Irinotecan, Capecitabine) (N=39)
Albumin, serum-low (hypoalbuminemia) (Blood and lymphatic system disorders) | 24
Alkaline phosphatase (Investigations) | 18
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 21
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 6
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 4
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 17
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 12
Diarrhea (Gastrointestinal disorders) | 29
Distension/bloating, abdominal (Gastrointestinal disorders) | 4
Dizziness (Nervous system disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 10
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9
Edema: limb (General disorders) | 6
Esophagitis (Gastrointestinal disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 29
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 5
Flushing (Vascular disorders) | 3
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 21
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Hemoglobin (Investigations) | 25
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Hot flashes/flushes (Vascular disorders) | 6
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Neck NOS (Infections and infestations) | 4
Infection with unknown ANC (Infections and infestations) | 4
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 2
Insomnia (Psychiatric disorders) | 11
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 18
Lymphopenia (Blood and lymphatic system disorders) | 15
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7
Mood alteration - Agitation (Psychiatric disorders) | 2
Mood alteration - Depression (Psychiatric disorders) | 4
Mucositis/stomatitis (Gastrointestinal disorders) | 7
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 10
Nausea (Gastrointestinal disorders) | 20
Neuropathy: sensory (Nervous system disorders) | 21
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14
Pain - Abdomen NOS (Gastrointestinal disorders) | 19
Pain - Back (Musculoskeletal and connective tissue disorders) | 9
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 5
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain - Head/headache (Nervous system disorders) | 3
Pain - Pain NOS (General disorders) | 4
Palpitations (Cardiac disorders) | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 3
Platelets (Blood and lymphatic system disorders) | 14
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 16
Proteinuria (Renal and urinary disorders) | 3
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
Rigors/chills (General disorders) | 2
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11
Supraventricular and nodal arrhythmia (Cardiac disorders) | 5
Sweating (diaphoresis) (Vascular disorders) | 3
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 3
Vision-blurred vision (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Weight gain (Investigations) | 3
Weight loss (Investigations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less